CLINICAL TRIAL: NCT01175135
Title: A Phase 2, Multicenter, Double-blind, Randomized, Parallel Group, 4-week Inpatient Study To Evaluate The Safety And Efficacy Of Two Fixed Doses Of Pf-02545920 Compared To Placebo In The Treatment Of Acute Exacerbation Of Schizophrenia Using Risperidone As An Active Control
Brief Title: An Inpatient Study Of The Efficacy, Safety, And Tolerability Of PF-02545920 In The Treatment Of Acute Exacerbation Of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A8241012; 2010-020764-38 (EudraCT Number)
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; acute exacerbation; inpatient
MeSH Terms: conditions — Schizophrenia | interventions — 2-((4-(1-methyl-4-pyridin-4-yl-1H-pyrazol-3-yl)phenoxy)methyl)quinoline; Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PF-02545920 5 mg (Experimental)
  Interventions: Drug: PF-02545920
- PF-02545920 15 mg (Experimental)
  Interventions: Drug: PF-02545920
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Risperidone 3 mg (Active Comparator)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: PF-02545920 — 5 mg tablet every 12 hours for 28 days
  Arms: PF-02545920 5 mg
Drug: PF-02545920 — 15 mg tablet every 12 hours for 28 days
  Arms: PF-02545920 15 mg
Drug: Placebo — One tablet/capsule every 12 hours for 28 days
  Arms: Placebo
Drug: Risperidone — 3 mg capsule every 12 hours for 28 days
  Other Names: Risperdal
  Arms: Risperidone 3 mg

SUMMARY:
This study aims to evaluate whether PF-02545920 is safe and effective in the treatment of acute exacerbation of schizophrenia during a 4-week inpatient treatment period. The study will use the Positive and Negative Syndrome Scale (PANSS) to measure change in symptoms for PF-02545920 compared to risperidone and placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia with acute exacerbation of illness
* The current acute exacerbation of schizophrenia must be less than 4 weeks duration prior to the initial evaluation.

Exclusion Criteria:

* Subjects with evidence or history of clinically significant uncontrolled medical illness
* Subjects with a current diagnosis of schizoaffective disorder, major depression, bipolar disorder, or obsessive compulsive disorder.
* Subjects who meet Diagnostic and Statistical Manual-IV (DSM-IV)defined diagnostic criteria for psychoactive substance dependence (excluding nicotine dependence) within 12 months of screening or DSM-IV defined substance abuse within 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- United States (38):
  - K & S Professional Research Services, LLC, Little Rock, Arkansas
  - Leisure Court Center, Anaheim, California
  - Early Phase Investigational Center, Escondido, California
  - Synergy Clinical Research Center of Escondido, Escondido, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Ocean View Psychiatric Health Facility, Long Beach, California
  - Long Beach VA Healthcare System, Long Beach, California
  - University of California Irvine Medical Center, Orange, California
  - California Clinical Trials Medical Group, Paramount, California
  - LaPaz Geropsychiatric Center, Paramount, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Collaborative Neuroscience Network, Inc., Torrance, California
  - Del Amo Hospital, Torrance, California
  - Comprehensive Neuroscience, Incorporated, Washington D.C., District of Columbia
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Lakeside Behavioral Healthcare, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Alexian Brothers Behavioral Health Hospital, Hoffman Estates, Illinois
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Chinmay K. Patel, D.O., Hoffman Estates, Illinois
  - Lake Charles Memorial Hospital, Lake Charles, Louisiana
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - CBH Health, LLC, Rockville, Maryland
  - St. Louis Clinical Trials, LC, St Louis, Missouri
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - Lourdes Medical Center of Burlington County, Willingboro, New Jersey
  - Comprehensive Neuroscience, Inc., Hollis, New York
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - FutureSearch Trials, Austin, Texas
  - TexasNeuroRehab Center, Austin, Texas
  - Community Clinical Research, Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Bayou City Research, Ltd., Houston, Texas
  - Behavioral Hospital - Bellaire, Houston, Texas
  - Eastside Therapeutic Resource, Kirkland, Washington
  - Fairfax Hospital, Kirkland, Washington
- Zentralinstitut fuer Seelische Gesundheit, Mannheim, Germany
- Ukraine (7):
  - Municipal Establishment "Dnipropetrovsk Regional Clinical Hospital n.a. Mechnikov", Dnipropetrovsk
  - Municipal Establishment "Dnipropetrovsk Regional Clinical Psychiatric Hospital", Dnipropetrovsk
  - Kyiv City Psychoneurological Hospital #2, Kyiv
  - Kyiv City Clinical Psychoneurological Hospital #1, Kyiv
  - Lugansk Regional Clinical Psychoneurological Hospital, Luhansk
  - Poltava Regional Clinical Psychiatric Hospital n.a. O.F. Maltsev, Poltava
  - Kherson Regional Psychiatric Hospital, Department #3, Stepanivka, Kherson

REFERENCES:
- [Derived] Targum SD, Little JA, Lopez E, Demartinis N, Rapaport M, Ereshefsky L. Application of external review for subject selection in a schizophrenia trial. J Clin Psychopharmacol. 2012 Apr;32(2):825-6. doi: 10.1097/JCP.0b013e318248da90. No abstract available. PMID 22388170
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8241012&StudyName=An%20Inpatient%20Study%20Of%20The%20Efficacy%2C%20Safety%2C%20And%20Tolerability%20Of%20PF-02545920%20In%20The%20Treatment%20Of%20Acute%20Exacerbation%20Of%20Schizophrenia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received placebo-matched to PF-02545920 tablet and placebo-matched to risperidone tablet-in-capsule orally every 12 hours for 2 days during the placebo lead-in phase (before randomization in the study).
Groups:
- PF-02545920 5 mg: Participants received PF-02545920 5 milligram (mg) tablet, orally every 12 hours for 28 days.
- PF-02545920 15 mg: Participants received PF-02545920 tablet, dose was titrated with a starting dose of 5 mg up to 15 mg, orally every 12 hours for 28 days.
- Risperidone 3 mg: Participants received risperidone tablet-in-capsule, dose was titrated with a starting dose of 1 mg up to 3 mg, orally every 12 hours for 28 days.
- Placebo: Participants received placebo-matched to PF-02545920 tablet and placebo-matched to risperidone tablet-in-capsule orally every 12 hours for 28 days.
Period: Overall Study
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Started | 74 | 74 | 37 | 74
Treated | 74 | 74 | 36 | 74
Analyzed for Efficacy | 74 | 73 | 34 | 73
Completed | 58 | 52 | 25 | 60
Not Completed | 16 | 22 | 12 | 14
Not completed — Adverse Event | 2 | 5 | 3 | 4
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 5 | 0 | 5
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 8 | 5 | 5
Not completed — Other | 3 | 1 | 3 | 0
Not completed — Randomized But Not Treated | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Included all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo | Total
Number analyzed (Participants) | 74 | 74 | 36 | 74 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (11.2) | 41.7 (10.5) | 41.3 (10.9) | 41.2 (10.9) | 41.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 11 | 18 | 60
  Male | 57 | 60 | 25 | 56 | 198

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 4
Description: PANSS assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210; higher score indicates greater severity.
Time Frame: Baseline, Week 4
Population: Full analysis set (FAS) included all participants who received at least 1 dose of randomized study medication, and had a baseline and at least 1 post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 73 | 34 | 73
units on a scale
  Baseline | 98.1 (11.81) | 97.7 (11.14) | 97.4 (15.05) | 97.2 (14.92)
  Change at Week 4: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4 | -15.3 (15.56) | -13.8 (17.93) | -17.9 (10.99) | -12.6 (15.29)
Statistical Analysis 1: Comparison: PF-02545920 5 mg vs Placebo; Mixed effect repeated measures (MMRM) model with fixed effect for baseline PANSS total score, investigator site, treatment, visit, treatment by visit interaction and baseline PANSS total score by visit interaction, and random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.2053, Mixed Models Analysis — Reported p-value was 1-sided; Least Squares (LS) Mean Difference = -2.21, 80% CI 2-sided [-5.66 to 1.24], Standard Error of Mean 2.683
Statistical Analysis 2: Comparison: PF-02545920 15 mg vs Placebo; MMRM model with fixed effect for baseline PANSS total score, investigator site, treatment, visit, treatment by visit interaction and baseline PANSS total score by visit interaction, and random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.4024, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.67, 80% CI 2-sided [-4.14 to 2.80], Standard Error of Mean 2.698
Statistical Analysis 3: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.0090, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -8.24, 80% CI 2-sided [-12.68 to -3.80], Standard Error of Mean 3.453

2. Primary Outcome: Proportion of Participants With Dystonia Adverse Events
Description: Participants were assessed for presence of symptoms for any one of the following: dystonia, oromandibular dystonia, and oculogyric crisis.
Time Frame: Baseline up to end of study (7 to 10 days after administration of last dose of study medication)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: proportion of participants
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 74 | 36 | 74
proportion of participants | 0.01 | 0.08 | 0.00 | 0.04
Statistical Analysis 1: Comparison: PF-02545920 5 mg vs Placebo; Test type: Other; Difference in Proportion = -0.03, 80% CI 2-sided [-0.07 to 0.01] — The adjusted 80% Confidence Interval (CI) equals 88.6% CI, adjusted due to 1 interim look
Statistical Analysis 2: Comparison: PF-02545920 15 mg vs Placebo; Test type: Other; Difference in Proportion = 0.04, 80% CI 2-sided [-0.02 to 0.10] — The adjusted 80% CI equals 88.6% CI, adjusted due to 1 interim look
Statistical Analysis 3: Comparison: Risperidone 3 mg vs Placebo; Test type: Other; Difference in Proportion = -0.04, 80% CI 2-sided [-0.08 to -0.00] — The adjusted 80% CI equals 88.6% CI, adjusted due to 1 interim look

3. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Positive, Negative, and General Subscales Score at Week 4
Description: PANSS - positive, negative, and general subscales assesses positive, negative and general psychopathological symptoms associated with schizophrenia respectively. Seven (7) items each make up the positive scale (for example; delusions, conceptual disorganization, and hallucinatory behavior) and negative scale (for example; blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal) and 16 items make up the general scale (for example; somatic concern, anxiety, guilt feelings, mannerisms and posturing, motor retardation, uncooperativeness, disorientation, poor impulse control, pre-occupation). Each item is rated on a 7-point Likert scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total scores range for positive as well as negative subscale is 7 to 49 and for general subscale is 16 to 112; higher subscale score indicates greater severity.
Time Frame: Baseline, Week 4
Population: FAS included all participants who received at least 1 dose of randomized study medication, and had a baseline and at least 1 post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 73 | 34 | 73
units on a scale
  Baseline: Positive Score | 26.9 (4.00) | 26.1 (3.89) | 26.6 (4.74) | 26.8 (4.16)
  Baseline: Negative Score | 23.4 (4.15) | 23.4 (4.32) | 24.0 (5.18) | 23.2 (5.12)
  Baseline: General Score | 47.9 (6.67) | 48.2 (6.43) | 46.8 (8.25) | 47.2 (7.73)
  Change at Week 4: Positive Score: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4: Positive Score | -5.0 (5.26) | -4.5 (5.51) | -6.7 (3.84) | -4.5 (4.68)
  Change at Week 4: Negative Score: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4: Negative Score | -2.7 (4.62) | -2.2 (5.09) | -2.7 (4.03) | -1.5 (3.78)
  Change at Week 4: General Score: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4: General Score | -7.5 (7.75) | -7.1 (8.80) | -8.6 (5.85) | -6.6 (8.20)
Statistical Analysis 1: Comparison: PF-02545920 5 mg vs Placebo; Positive Score: MMRM model with fixed effect for baseline PANSS positive subscale score, investigator site, treatment, visit, a treatment by visit interaction and a baseline PANSS positive subscale score by visit interaction and a random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.3144, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.41, 80% CI 2-sided [-1.50 to 0.68], Standard Error of Mean 0.845
Statistical Analysis 2: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.5700, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = 0.15, 80% CI 2-sided [-0.95 to 1.25], Standard Error of Mean 0.854
Statistical Analysis 3: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.0034, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -2.99, 80% CI 2-sided [-4.40 to -1.59], Standard Error of Mean 1.093
Statistical Analysis 4: Comparison: PF-02545920 5 mg vs Placebo; Negative Score: MMRM model with fixed effect for baseline PANSS negative subscale score, investigator site, treatment, visit, a treatment by visit interaction and a baseline PANSS negative subscale score by visit interaction and a random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.0942, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.96, 80% CI 2-sided [-1.90 to -0.02], Standard Error of Mean 0.730
Statistical Analysis 5: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Other; p = 0.2030, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.61, 80% CI 2-sided [-1.56 to 0.33], Standard Error of Mean 0.735
Statistical Analysis 6: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Other; p = 0.0907, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -1.26, 80% CI 2-sided [-2.48 to -0.05], Standard Error of Mean 0.944
Statistical Analysis 7: Comparison: PF-02545920 5 mg vs Placebo; General Score: MMRM model with fixed effect for baseline PANSS general subscale score, investigator site, treatment, visit, a treatment by visit interaction and a baseline PANSS general subscale score by visit interaction and a random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.2904, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.74, 80% CI 2-sided [-2.45 to 0.97], Standard Error of Mean 1.330
Statistical Analysis 8: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Other; p = 0.4710, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.10, 80% CI 2-sided [-1.82 to 1.62], Standard Error of Mean 1.339
Statistical Analysis 9: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Other; p = 0.0172, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -3.66, 80% CI 2-sided [-5.86 to -1.45], Standard Error of Mean 1.718

4. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Week 4
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state. Clinician responded to a question "Considering your total clinical experience with this particular population, how mentally ill is your patient at this time?" on the following scores: 1 (normal - not ill at all), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill), 7 (among the most severely ill participants). Higher score = more affected.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 73 | 34 | 73
units on a scale
  Baseline | 5.0 (0.56) | 5.0 (0.49) | 4.9 (0.67) | 5.0 (0.58)
  Change at Week 4: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4 | -0.7 (0.87) | -0.7 (1.06) | -0.8 (0.78) | -0.6 (0.92)
Statistical Analysis 1: Comparison: PF-02545920 5 mg vs Placebo; MMRM model with fixed effect for baseline CGI-S, investigator site, treatment, visit, treatment by visit interaction, a baseline CGI-S by visit interaction and random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.1970, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.13, 80% CI 2-sided [-0.33 to 0.07], Standard Error of Mean 0.154
Statistical Analysis 2: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.3835, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.05, 80% CI 2-sided [-0.24 to 0.15], Standard Error of Mean 0.154
Statistical Analysis 3: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.0395, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.35, 80% CI 2-sided [-0.61 to -0.10], Standard Error of Mean 0.199

5. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Marder Factors Score at Week 4
Description: PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). PANSS Marder positive symptoms subscale consists of 8 items with total score equal to sum of 8 items ranging from 8-56; Marder negative symptoms subscale and Marder disorganized thoughts (Dis. Thought) subscale, each consists of 7 items with total score equal to sum of 7 items each, ranging from 7-49, Marder uncontrolled hostility/excitement (Uncon. Hos/Exc) subscale and Marder anxiety/depression (Anx/Dep) subscale, each consists of 4 items with total score equal to sum of 4 items each ranging from 4-28. Higher subscale score indicates greater severity.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 73 | 34 | 73
units on a scale
  Baseline: Positive score | 30.9 (4.51) | 30.6 (4.12) | 30.3 (5.45) | 31.0 (4.68)
  Baseline: Negative Score | 23.0 (4.43) | 23.3 (4.99) | 22.9 (5.04) | 23.0 (5.06)
  Baseline: Dis. Thought Score | 20.4 (5.13) | 21.0 (4.37) | 21.3 (5.49) | 20.3 (5.70)
  Baseline: Uncon. Hos/Exc Score | 10.4 (2.92) | 9.8 (2.98) | 10.6 (3.97) | 10.0 (3.44)
  Baseline: Anx/Dep Score | 13.5 (2.81) | 13.0 (3.16) | 12.4 (3.17) | 12.9 (2.56)
  Change at Week 4: Positive score: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4: Positive score | -5.5 (5.34) | -5.0 (5.56) | -6.2 (4.53) | -4.6 (5.00)
  Change at Week 4: Negative Score: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4: Negative Score | -3.0 (4.99) | -2.9 (5.69) | -2.5 (4.44) | -2.3 (4.91)
  Change at Week 4:Dis. Thought Score: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4:Dis. Thought Score | -2.5 (3.47) | -2.3 (4.39) | -3.0 (3.06) | -1.9 (3.05)
  Change at Week 4:Uncon.Hos/ExcScore: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4:Uncon.Hos/ExcScore | -1.2 (3.31) | -0.9 (3.12) | -2.4 (2.28) | -1.0 (2.95)
  Change at Week 4: Anx/DepScore: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4: Anx/DepScore | -2.9 (3.72) | -2.6 (3.85) | -3.8 (3.31) | -2.9 (3.22)
Statistical Analysis 1: Comparison: PF-02545920 5 mg vs Placebo; Positive Score: MMRM model with fixed effect for baseline PANSS Marder positive score, investigator site, treatment, visit, treatment by visit interaction and baseline PANSS Marder positive score by visit interaction, and random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.1999, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.73, 80% CI 2-sided [-1.84 to 0.38], Standard Error of Mean 0.863
Statistical Analysis 2: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.3399, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.36, 80% CI 2-sided [-1.48 to 0.76], Standard Error of Mean 0.870
Statistical Analysis 3: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.0100, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -2.62, 80% CI 2-sided [-4.06 to -1.18], Standard Error of Mean 1.117
Statistical Analysis 4: Comparison: PF-02545920 5 mg vs Placebo; Negative Score: MMRM model with fixed effect for baseline PANSS Marder negative score, investigator site, treatment, visit, treatment by visit interaction and baseline PANSS Marder negative score by visit interaction, and random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.1625, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.77, 80% CI 2-sided [-1.77 to 0.23], Standard Error of Mean 0.778
Statistical Analysis 5: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 5, analysis 4]; Test type: Other; p = 0.2354, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.57, 80% CI 2-sided [-1.57 to 0.44], Standard Error of Mean 0.783
Statistical Analysis 6: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 5, analysis 4]; Test type: Other; p = 0.2161, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.79, 80% CI 2-sided [-2.08 to 0.50], Standard Error of Mean 1.002
Statistical Analysis 7: Comparison: PF-02545920 5 mg vs Placebo; Disorganized Thought Score: MMRM model with fixed effect for baseline PANSS Marder disorganized thought score, investigator site, treatment, visit, treatment by visit interaction and baseline PANSS Marder disorganized thought score by visit interaction, and random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.2480, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.43, 80% CI 2-sided [-1.23 to 0.38], Standard Error of Mean 0.627
Statistical Analysis 8: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Other; p = 0.4345, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.10, 80% CI 2-sided [-0.92 to 0.71], Standard Error of Mean 0.632
Statistical Analysis 9: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Other; p = 0.0346, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -1.48, 80% CI 2-sided [-2.53 to -0.44], Standard Error of Mean 0.813
Statistical Analysis 10: Comparison: PF-02545920 5 mg vs Placebo; Uncontrolled hostility/excitement Score: MMRM model with fixed effect for baseline PANSS Marder hostility/excitement score, investigator site, treatment, visit, treatment by visit interaction and baseline PANSS Marder hostility/excitement score by visit interaction, and random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.4685, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.04, 80% CI 2-sided [-0.68 to 0.60], Standard Error of Mean 0.495
Statistical Analysis 11: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 5, analysis 10]; Test type: Other; p = 0.6214, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = 0.15, 80% CI 2-sided [-0.49 to 0.80], Standard Error of Mean 0.499
Statistical Analysis 12: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 5, analysis 10]; Test type: Other; p = 0.0052, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -1.66, 80% CI 2-sided [-2.48 to -0.84], Standard Error of Mean 0.641
Statistical Analysis 13: Comparison: PF-02545920 5 mg vs Placebo; Anxiety/Depression Score: MMRM model with fixed effect for baseline PANSS Marder anxiety/depression score, investigator site, treatment, visit, treatment by visit interaction and baseline PANSS Marder anxiety/depression score by visit interaction, and random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.5894, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = 0.12, 80% CI 2-sided [-0.55 to 0.79], Standard Error of Mean 0.523
Statistical Analysis 14: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 5, analysis 13]; Test type: Other; p = 0.8155, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = 0.47, 80% CI 2-sided [-0.20 to 1.15], Standard Error of Mean 0.526
Statistical Analysis 15: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 5, analysis 13]; Test type: Other; p = 0.0069, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -1.68, 80% CI 2-sided [-2.55 to -0.81], Standard Error of Mean 0.677

6. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Derived Brief Psychiatric Rating Scale (BPRS) Core Score at Week 4
Description: PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. PANSS derived BPRS is an 18-item clinician rated scale which assesses symptoms such as hostility, suspiciousness, hallucinations, grandiosity, and a number of other psychiatric symptoms. Items scored on a 7-point scale (1=not present and 7=extremely severe), with higher score indicating greater severity of symptom. BPRS core score consists of 4 items (Conceptual disorganization, Hallucinatory behavior, Suspiciousness/persecution, Unusual thought content) with total score equal to sum of the 4 items, ranging from 4 to 28, with higher score indicating greater severity.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 73 | 34 | 73
units on a scale
  Baseline | 17.4 (2.74) | 17.3 (2.32) | 17.2 (2.77) | 17.3 (2.39)
  Change at Week 4: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4 | -3.7 (3.39) | -3.4 (3.75) | -4.7 (2.99) | -3.2 (3.12)
Statistical Analysis 1: Comparison: PF-02545920 5 mg vs Placebo; MMRM model with fixed effect for baseline PANSS derived BPRS core score, investigator site, treatment, visit, treatment by visit interaction and baseline PANSS derived BPRS core score by visit interaction, and random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.2727, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.34, 80% CI 2-sided [-1.06 to 0.38], Standard Error of Mean 0.559
Statistical Analysis 2: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.4747, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.04, 80% CI 2-sided [-0.76 to 0.69], Standard Error of Mean 0.562
Statistical Analysis 3: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.0031, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -2.00, 80% CI 2-sided [-2.93 to -1.07], Standard Error of Mean 0.723

7. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Score
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Clinician responded to a question: "Compared to your subject's condition at the beginning of treatment, how much has your subject changed?" Compared to Baseline (Day 1), improvement was defined as score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 63 | 58 | 26 | 63
units on a scale | 3.1 (0.98) | 3.3 (1.35) | 2.7 (0.89) | 3.2 (1.05)
Statistical Analysis 1: Comparison: PF-02545920 5 mg vs Placebo; MMRM model with fixed effect for investigator site, treatment, visit, treatment by visit interaction and random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.3598, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.07, 80% CI 2-sided [-0.32 to 0.18], Standard Error of Mean 0.196
Statistical Analysis 2: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.7275, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = 0.12, 80% CI 2-sided [-0.13 to 0.37], Standard Error of Mean 0.198
Statistical Analysis 3: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0019, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.75, 80% CI 2-sided [-1.07 to -0.42], Standard Error of Mean 0.255

8. Secondary Outcome: Change From Baseline in Global Assessment of Functioning (GAF) Score at Week 4
Description: GAF is a 100-point, clinician rated single item scale that rates the severity of illness-related impairment in psychological, social and occupational functioning of participants on a hypothetical continuum of mental illness to mental health. The scale values range from 1 to 100 with lower score indicating greater severity of illness and is divided into 10 equal intervals (descriptors): from 1-10 (persistent danger of hurting self - serious suicidal acting with clear expectations of death) to 91-100 (superior functioning - no symptoms). Each descriptor has a nine-point range to allow for some variability of severity within the descriptor.
Time Frame: Baseline, Week 4
Population: FAS. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 73 | 71 | 34 | 72
units on a scale
  Baseline | 38.4 (8.31) | 38.5 (7.82) | 38.7 (10.58) | 38.2 (8.78)
  Change at Week 4: number analyzed (Participants) | 62 | 57 | 26 | 62
  Change at Week 4 | 6.3 (9.08) | 6.9 (8.92) | 7.7 (8.45) | 6.3 (8.14)
Statistical Analysis 1: Comparison: PF-02545920 5 mg vs Placebo; MMRM model with fixed effect for baseline GAF score, investigator site, treatment, visit, treatment by visit interaction, baseline GAF score by visit interaction and random effect for participant. The model was fit using an unstructured covariance matrix; Test type: Other; p = 0.5429, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = -0.16, 80% CI 2-sided [-2.06 to 1.74], Standard Error of Mean 1.478
Statistical Analysis 2: Comparison: PF-02545920 15 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.4354, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = 0.24, 80% CI 2-sided [-1.68 to 2.16], Standard Error of Mean 1.492
Statistical Analysis 3: Comparison: Risperidone 3 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.0930, Mixed Models Analysis — Reported p-value was 1-sided; LS Mean Difference = 2.53, 80% CI 2-sided [0.08 to 4.99], Standard Error of Mean 1.907

9. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) Score
Description: TSQM assesses the participant's level of satisfaction with study medication. It consists of a 14-item questionnaire which comprises of 3 specific scales (effectiveness, side effects, convenience) and 1 global satisfaction scale. Effectiveness, convenience and global satisfaction scale are rated on a 7-point scale (0= Extremely Dissatisfied, 1= Very Dissatisfied, 2= Dissatisfied, 3= Somewhat Satisfied, 4= Satisfied, 5= Very Satisfied, 6= Extremely Satisfied) and side effects are rated on a 5-point scale (0= Extremely Dissatisfied, 1=Very Dissatisfied, 2= Somewhat Dissatisfied, 3= Slightly Dissatisfied, 4= Not at all Dissatisfied). Scale scores are transformed into scores ranging from 0 to 100, with a higher score indicating more satisfaction.
Time Frame: Week 4
Population: FAS. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 71 | 70 | 32 | 69
units on a scale
  Effectiveness | 53.68 (24.84) | 51.90 (24.28) | 63.37 (24.07) | 53.70 (19.68)
  Side-Effects: number analyzed (Participants) | 70 | 70 | 32 | 69
  Side-Effects | 86.43 (24.45) | 79.20 (28.67) | 87.30 (22.02) | 87.41 (24.00)
  Convenience | 70.46 (17.46) | 68.37 (18.49) | 75.69 (15.44) | 66.83 (15.12)
  Global Satisfaction | 56.84 (28.30) | 51.02 (27.79) | 66.07 (23.38) | 49.48 (24.69)

10. Secondary Outcome: Change From Baseline in Body Weight at Week 4
Time Frame: Baseline, Week 4
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 72 | 36 | 74
kilogram (kg)
  Baseline | 86.1 (15.06) | 87.5 (14.46) | 83.9 (16.99) | 84.3 (19.31)
  Change at Week 4: number analyzed (Participants) | 72 | 69 | 32 | 70
  Change at Week 4 | 0.18 (2.23) | -1.23 (3.18) | 2.69 (3.00) | 1.04 (2.61)

11. Secondary Outcome: Change From Baseline in Abdominal Girth at Week 4
Time Frame: Baseline, Week 4
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 72 | 36 | 72
centimeter (cm)
  Baseline | 96.5 (12.33) | 97.2 (13.49) | 95.6 (13.58) | 93.5 (16.05)
  Change at Week 4: number analyzed (Participants) | 72 | 69 | 32 | 68
  Change at Week 4 | 0.71 (5.07) | 0.70 (5.73) | 3.33 (4.54) | 0.74 (4.29)

12. Secondary Outcome: Number of Participants With Clinically Significant Findings in Vital Signs and Electrocardiogram (ECG)
Description: Clinically significant findings based on investigator's discretion were assessed in vital sign parameters (including pulse rate, blood pressure and body temperature) and ECG parameters (including respiratory rate, heart rate, PR interval, QRS interval, QT interval, QT corrected using Bazett's correction [QTcB] interval, and QT corrected using Fridericia's correction [QTcF]).
Time Frame: Baseline up to end of study (7 to 10 days after administration of last dose of study medication)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 74 | 36 | 74
participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Physical Examinations
Description: Clinically significant findings in physical examinations based on investigator's discretion were assessed. Screening was the 7 day time (from Day -8 to Day -2) before dosing on Day 1. Number of participants with clinically significant changes in physical examinations compared to screening was assessed.
Time Frame: Screening, Week 4
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 74 | 36 | 74
participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for abnormality:hematology: hemoglobin, hematocrit, red blood cell count: less than(<) 0.8*lower limit of normal (LLN); mean corpuscular volume; mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration: <0.9*LLN,>1.1*upper limit of normal (ULN); platelets: <0.5*LLN,>1.75*ULN, white blood cell count: <0.6*LLN, >1.5*ULN; lymphocytes, total neutrophils: <0.8*LLN, >1.2*ULN; eosinophils, basophils, monocytes: >1.2*ULN; coagulation: activated partial thromboplastin time, prothrombin, prothrombin international ratio: >1.1*ULN; liver function: bilirubin: >1.5*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase: >3.0*ULN; protein, albumin: <0.8*LLN></0>1.2*ULN; renal function:blood urea nitrogen,creatinine: >1.3*ULN; uric acid: >1.2*ULN; electrolytes: sodium, potassium, chloride, calcium, bicarbonate: <0.9*LLN,>1.1*ULN; urinalysis: pH<4.5, >8; glucose, protein, blood, ketones, urobilinogen, bilirubin, nitrite; Other(glucose: <0.6*LLN,>1.5*ULN)
Time Frame: Screening up to end of study (7 to 10 days after administration of last dose of study medication)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 74 | 35 | 74
participants | 55 | 58 | 34 | 56

15. Secondary Outcome: Number of Participants With Abnormal White Blood Cell (WBC) Count and Absolute Neutrophil Count (ANC)
Description: Pre-defined criteria was established for WBC Count (less than 0.6 times the lower limit of normal) and absolute neutrophil count (less than 0.8 times the lower limit of normal) to define the values that would be identified as abnormal.
Time Frame: Day 1 up to Week 4
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 74 | 35 | 74
participants
  WBC | 0 | 0 | 0 | 0
  ANC | 6 | 6 | 0 | 8

16. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities for Fasting Insulin, High Density Lipoprotein (HDL), Low Density Lipoprotein (LDL), Cholesterol, Triglycerides, Hemoglobin Type A1c (HbA1c) and Prolactin
Description: Clinically significant findings based on investigator's discretion were assessed in laboratory parameters (including fasting insulin, high-density lipoprotein [HDL], low-density lipoprotein [LDL], Cholesterol, Triglycerides, glycosylated hemoglobin type A1c [HbA1c] and Prolactin).
Time Frame: Day 1 up to Week 4
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 74 | 35 | 74
participants | 0 | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline in Extrapyramidal Symptom Rating Scale-Abbreviated (ESRS-A) Parameter Scores at Week 4
Description: ESRS-A is a clinician rated scale consisting of 24 items to assess severity of extra-pyramidal symptoms for following parameters: parkinsonism (10 items), dystonia (6 items), dyskinesia (6 items) and akathisia (2 items). Each item is scored on a 6-point Likert scale (0=absent, 1=minimal, 2=mild, 3=moderate, 4=severe, 5=extreme). Total score for a parameter is average of individual item scores included under the parameter, ranging from 0 to 5, with higher score = more affected.
Time Frame: Baseline, Week 4
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 74 | 36 | 74
units on a scale
  Baseline: Parkinsonism | 0.257 (1.0476) | 0.500 (1.5283) | 0.194 (0.6242) | 0.473 (1.5809)
  Baseline: Dystonia | 0.095 (0.5278) | 0.000 (0.0000) | 0.000 (0.0000) | 0.027 (0.1633)
  Baseline: Dyskinesia | 0.122 (0.4038) | 0.095 (0.4432) | 0.194 (0.5767) | 0.135 (0.5054)
  Baseline: Akathisia | 0.162 (0.5496) | 0.068 (0.4778) | 0.111 (0.6667) | 0.243 (0.7551)
  Change at Week 4: Parkinsonism: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4: Parkinsonism | 0.143 (0.8397) | 0.086 (1.3414) | -0.038 (0.9157) | -0.190 (1.4126)
  Change at Week 4: Dystonia: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4: Dystonia | 0.000 (0.4016) | 0.207 (1.1044) | 0.000 (0.0000) | 0.032 (0.2520)
  Change at Week 4: Dyskinesia: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4: Dyskinesia | 0.016 (0.4916) | 0.207 (1.0884) | 0.038 (0.4455) | -0.032 (0.3578)
  Change at Week 4: Akathisia: number analyzed (Participants) | 63 | 58 | 26 | 63
  Change at Week 4: Akathisia | 0.032 (0.6713) | 0.328 (1.3297) | 0.154 (1.2866) | -0.095 (0.9283)

18. Secondary Outcome: Change From Baseline in Movement Disorder Burden Score for Dystonia (MDBS-D) at Week 4
Description: MDBS-D score reflects the numbers and durations of movement disorder adverse events for dystonia, the severity of the events, required treatment, and the total number of days the participant received study treatment. MDBS-D score = (S * D * C)/TTD; where S= Movement Disorder Severity Score for Dystonia (possible values: 1 [mild]; 2 [moderate]; 3 [severe]), D=adverse event duration (in days), C=concomitant medication factor (C=1.5 if an anti-cholinergic or beta blocker is used for the treatment of a movement disorder; C=1 if no concomitant medication is used), TTD=total treatment days for the participant. Value for MDBS score may range from zero to infinity. A higher MDBS-D score indicates a greater movement disorder adverse event liability compared to baseline.
Time Frame: Baseline, Week 4
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 74 | 36 | 74
units on a scale | 0.0019 (0.01648) | 0.0163 (0.08087) | 0.0000 (0.00000) | 0.0126 (0.10349)

19. Secondary Outcome: Number of Participants With Response to Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Data relevant to the assessment of suicidality is mapped to the Columbia Classification Algorithm of Suicide Assessment (C-CASA) event codes. C-SSRS assesses whether participant experiences following: suicide attempt (Event code 2) (Response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (Event code 3) ("Yes" on "aborted attempt", "interrupted attempt", "preparatory acts or behavior"), suicidal ideation (Event code 4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act/some intent to act without specific plan or with specific plan and intent), self-injurious behavior, no suicidal intent (Event code 7) ("Yes" on "Has participant engaged in non-suicidal self-injurious behavior"). Number of participants with "Yes" response for above mentioned categories are assessed. Baseline is defined as the Week 0 measurement.
Time Frame: Baseline, Week 1, 2, 3, 4, Follow-up (FU) (7 to 10 days after administration of last dose of study medication)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Number analyzed (Participants) | 74 | 74 | 36 | 74
participants
  Baseline: Event code 2 | 1 | 1 | 0 | 1
  Baseline: Event code 3 | 1 | 0 | 0 | 2
  Baseline: Event code 4 | 1 | 4 | 1 | 3
  Baseline: Event code 7 | 0 | 1 | 0 | 0
  Week 1: Event code 2: number analyzed (Participants) | 74 | 74 | 34 | 73
  Week 1: Event code 2 | 0 | 0 | 0 | 0
  Week 1: Event code 3: number analyzed (Participants) | 74 | 74 | 34 | 73
  Week 1: Event code 3 | 0 | 1 | 0 | 0
  Week 1: Event code 4: number analyzed (Participants) | 74 | 74 | 34 | 73
  Week 1: Event code 4 | 0 | 4 | 0 | 0
  Week 1: Event code 7: number analyzed (Participants) | 74 | 74 | 34 | 73
  Week 1: Event code 7 | 0 | 0 | 0 | 0
  Week 2: Event code 2: number analyzed (Participants) | 71 | 72 | 32 | 69
  Week 2: Event code 2 | 0 | 0 | 0 | 0
  Week 2: Event code 3: number analyzed (Participants) | 71 | 72 | 32 | 69
  Week 2: Event code 3 | 0 | 0 | 0 | 0
  Week 2: Event code 4: number analyzed (Participants) | 71 | 72 | 32 | 69
  Week 2: Event code 4 | 1 | 3 | 0 | 1
  Week 2: Event code 7: number analyzed (Participants) | 71 | 72 | 32 | 69
  Week 2: Event code 7 | 0 | 0 | 0 | 0
  Week 3: Event code 2: number analyzed (Participants) | 68 | 69 | 28 | 69
  Week 3: Event code 2 | 0 | 0 | 0 | 0
  Week 3: Event code 3: number analyzed (Participants) | 68 | 69 | 28 | 69
  Week 3: Event code 3 | 0 | 0 | 0 | 0
  Week 3: Event code 4: number analyzed (Participants) | 68 | 69 | 28 | 69
  Week 3: Event code 4 | 0 | 2 | 0 | 1
  Week 3: Event code 7: number analyzed (Participants) | 68 | 69 | 28 | 69
  Week 3: Event code 7 | 0 | 0 | 0 | 0
  Week 4: Event code 2: number analyzed (Participants) | 66 | 63 | 27 | 64
  Week 4: Event code 2 | 0 | 0 | 0 | 0
  Week 4: Event code 3: number analyzed (Participants) | 66 | 63 | 27 | 64
  Week 4: Event code 3 | 0 | 0 | 0 | 0
  Week 4: Event code 4: number analyzed (Participants) | 66 | 63 | 27 | 64
  Week 4: Event code 4 | 3 | 3 | 1 | 0
  Week 4: Event code 7: number analyzed (Participants) | 66 | 63 | 27 | 64
  Week 4: Event code 7 | 0 | 0 | 0 | 0
  FU: Event code 2: number analyzed (Participants) | 61 | 53 | 26 | 63
  FU: Event code 2 | 0 | 0 | 0 | 0
  FU: Event code 3: number analyzed (Participants) | 61 | 53 | 26 | 63
  FU: Event code 3 | 0 | 0 | 0 | 0
  FU: Event code 4: number analyzed (Participants) | 61 | 53 | 26 | 63
  FU: Event code 4 | 1 | 0 | 1 | 0
  FU: Event code 7: number analyzed (Participants) | 61 | 53 | 26 | 63
  FU: Event code 7 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-02545920 5 mg | PF-02545920 15 mg | Risperidone 3 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/74 | 6/74 | 2/36 | 1/74
Other Adverse Events (participants affected / at risk) | 53/74 | 47/74 | 22/36 | 51/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02545920 5 mg (N=74) | PF-02545920 15 mg (N=74) | Risperidone 3 mg (N=36) | Placebo (N=74)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial rupture (Cardiac disorders) | 1 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 2 | 0 | 1
Schizophrenia (Psychiatric disorders) | 1 | 3 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02545920 5 mg (N=74) | PF-02545920 15 mg (N=74) | Risperidone 3 mg (N=36) | Placebo (N=74)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 2 | 1 | 4
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 3 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 2 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Oculogyric crisis (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 8 | 2 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 1 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 3 | 6
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 6 | 3 | 5
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Toothache (Gastrointestinal disorders) | 2 | 2 | 1 | 4
Vomiting (Gastrointestinal disorders) | 2 | 3 | 2 | 5
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Feeling jittery (General disorders) | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 1 | 2
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 1
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0
Infected bites (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 2
Otitis media (Infections and infestations) | 0 | 0 | 0 | 2
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 2
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Blood insulin increased (Investigations) | 0 | 0 | 1 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 2 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Nuchal rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 0
Akathisia (Nervous system disorders) | 6 | 5 | 1 | 1
Aphonia (Nervous system disorders) | 1 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 0 | 4
Drooling (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1 | 0 | 0
Dystonia (Nervous system disorders) | 0 | 3 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 2 | 1 | 0 | 1
Headache (Nervous system disorders) | 15 | 10 | 9 | 11
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Movement disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Oromandibular dystonia (Nervous system disorders) | 1 | 2 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 1 | 0 | 0
Sedation (Nervous system disorders) | 3 | 5 | 1 | 3
Somnolence (Nervous system disorders) | 2 | 4 | 1 | 2
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 2 | 2 | 1 | 2
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 2 | 1 | 1
Delusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 3 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 2 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 2 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1 | 0
Enuresis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Galactorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.